CLINICAL TRIAL: NCT02204748
Title: Kinematic Analysis: Posterior Stabilized, Fixed Bearing Total Knee Arthroplasty
Brief Title: Kinematic Analysis: Posterior Stabilized, Fixed Bearing Total Knee Arthroplasty With Attune Knee System
Status: Completed | Type: Observational
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: DePuy Orthopaedics (Industry)
Responsible Party: Principal Investigator, Richard Komistek, Principal Investigator, The University of Tennessee, Knoxville
Other Study IDs: 13002; R011373503 (Other: University of Tennessee)
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Results first posted 2016-02-04 (Estimated); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Total Knee Arthroplasty; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DePuy Attune PS FB TKA: Individuals implanted with the DePuy Attune posterior stabilizing fixed bearing knee system implanted by a single surgeon at least three months post-operative.
  Interventions: Device: DePuy Attune posterior stabilizing fixed bearing knee system

INTERVENTIONS:
Device: DePuy Attune posterior stabilizing fixed bearing knee system

SUMMARY:
A better understanding of knee joint kinematics is important to explain the premature polyethylene wear failures within total knee arthroplasties (TKAs) and to help design a prosthesis that most closely approximates the normal knee. Specifically, posterior stabilizing (PS) knees have been found to be associated with lower amounts of posterior femoral rollback, higher occurrence of reverse axial rotation and increased amount of condylar lift-off. The DePuy Synthes Joint Reconstruction's Attune PS fixed bearing (FB) knee system has incorporated subtle changes in its design to address restoration of kinematics that more closely resemble those of a normal knee. To understand if this design is able to effectively restore kinematics in the implanted knee, further in vivo analysis is necessary. This pilot study will analyze 5 subjects with the Attune PS FB 3 months post-operatively using the University of Tennessee's mobile fluoroscopy unit while performing three daily activities, level walking, ramp down and deep knee bend. Since this is a pilot study, there is no hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* At least three (3) months post-operative with no other surgical procedures conducted within the past six months
* Between 30-80 years of age
* Body weight of less than 280 lbs
* Must be between 160cm (5'3) and 193cm (6'4) tall
* Body Mass Index (BMI) >18.5 and <35
* Judged clinically successful with a Knee Society score (KSS) of greater than 80
* Have good-to-excellent post-operative passive flexion with no ligamentous laxity or pain
* Must be able to walk on level ground without aid of any kind, perform a ramp descent, and a deep knee bend (DKB), all without assistance
* Will have a DePuy Attune PS TKA
* Must be willing to sign the Informed Consent (IC) and HIPAA forms to participate in the study

Exclusion Criteria:

- Pregnant or potentially pregnant females will be excluded from the study

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will have been implanted with the DePuy Attune PS FB knee system by Dr. Thomas Fehring of OrthoCarolina, PA in Charlotte, NC.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2014-11; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrija Sharma, Ph. D., Principal Investigator — University of Tennessee; William R Hamel, Ph. D., Principal Investigator — University of Tennessee
Locations (2):
- United States (2):
  - OrthoCarolina Research Institute, Charlotte, North Carolina
  - The University of Tennessee, Knoxville, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- DePuy Attune PS FB TKA: Individuals implanted with the DePuy Attune posterior stabilizing fixed bearing knee system implanted by a single surgeon at least three months post-operative.
  DePuy Attune posterior stabilizing fixed bearing knee system
Period: Overall Study
Arm/Group | DePuy Attune PS FB TKA
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | DePuy Attune PS FB TKA
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (8.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Femoro-tibial Kinematics - Translation and Lift-off for Deep Knee Bend
Description: Amount of translation and lift-off for implanted knee in vivo under fluoroscopic surveillance during deep knee bend activity.
Time Frame: 3 months post-operative
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | DePuy Attune PS FB TKA
Number analyzed (Participants) | 5
mm
  Lateral Anterior Posterior Deep Knee Bend | -4.89 (3.57)
  Medial Anterior Posterior Deep Knee Bend | -2.58 (2.5)

2. Primary Outcome: Femoro-tibial Kinematics: Translation and Lift-off for Gait
Description: Amount of translation and lift-off for implanted knee in vivo under fluoroscopic surveillance during gait activity.
Time Frame: 3 months post-operative
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | DePuy Attune PS FB TKA
Number analyzed (Participants) | 5
mm
  Lateral Anterior Posterior Gait | -0.8 (1.89)
  Medial Anterior Posterior Gait | 0.24 (0.67)

3. Primary Outcome: Femoro-tibial Kinematics: Translation and Lift-off for Ramp Down
Description: Amount of translation and lift-off for implanted knee in vivo under fluoroscopic surveillance during ramp down activity.
Time Frame: 3 months post-operative
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | DePuy Attune PS FB TKA
Number analyzed (Participants) | 5
mm
  Lateral Anterior Posterior Ramp Down | -1.35 (2.39)
  Medial Anterior Posterior Ramp Down | -0.58 (1.72)

4. Secondary Outcome: Max Ground Reaction Force - Deep Knee Bend
Description: Collected simultaneously with fluoroscopy data, ground reaction forces were obtained using a force plate (fixed to the ground) while subject performed activity. Maximum force measured in the vertical direction measured during the described activity, then normalized with respect to participant's body weight. As such, the data are presented as the percentage of the individuals' body weight that was supported on the implanted knee using a force plate (fixed to the ground) and has been termed "maximum reaction force."
Time Frame: 3 months post-operative
Measure: Mean (Standard Deviation); unit: percentage of body weight
Arm/Group | DePuy Attune PS FB TKA
Number analyzed (Participants) | 5
percentage of body weight | 75.3 (11.2)

5. Secondary Outcome: Max Ground Reaction Force - Gait
Description: as for outcome 4
Time Frame: 3 months post-operative
Measure: Mean (Standard Deviation); unit: percentage of body weight
Arm/Group | DePuy Attune PS FB TKA
Number analyzed (Participants) | 5
percentage of body weight | 106.0 (3.0)

6. Secondary Outcome: Max Ground Reaction Force - Ramp Down
Description: Collected simultaneously with fluoroscopy data, ground reaction forces were obtained using a force plate (fixed to the ground) while subject performed activity. Maximum force measured in the vertical direction measured during the described activity was normalized with respect to participant's body weight. As such, the data are presented as the percentage of the individuals' body weight that was supported on the implanted knee using a force plate (fixed to the ground) and has been termed "maximum reaction force."
Time Frame: 3 months post-operative
Measure: Mean (Standard Deviation); unit: percentage of body weight
Arm/Group | DePuy Attune PS FB TKA
Number analyzed (Participants) | 5
percentage of body weight | 97.2 (15.0)

7. Primary Outcome: Femoro-tibial Kinematics - Deep Knee Bend
Description: Degree of axial rotation and weight-bearing range-of-motion for implanted knee in vivo under fluoroscopic surveillance during deep knee bend activity.
Time Frame: 3 months post-operative
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | DePuy Attune PS FB TKA
Number analyzed (Participants) | 5
degrees
  Axial Rotation Deep Knee Bend | 2.99 (5.73)
  Max weight-bearing flexion Deep knee bend | 118.2 (20.96)

8. Primary Outcome: Femoro-tibial Kinematics - Gait
Description: Degree of axial rotation and weight-bearing range-of-motion for implanted knee in vivo under fluoroscopic surveillance during gait activity.
Time Frame: 3 months post-operative
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | DePuy Attune PS FB TKA
Number analyzed (Participants) | 5
degrees
  Axial Rotation Gait | 1.28 (2.76)
  Max Weight-bearing flexion Gait | 19.4 (4.72)

9. Primary Outcome: Femoro-tibial Kinematics - Ramp Down
Description: Degree of axial rotation and maximum weight-bearing range-of-motion for implanted knee in vivo under fluoroscopic surveillance during ramp down activity.
Time Frame: 3 months post-operative
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | DePuy Attune PS FB TKA
Number analyzed (Participants) | 5
degrees
  Axial Rotation Ramp Down | 0.97 (4.32)
  Max Weight-bearing flexion Ramp Down | 28.6 (5.94)

ADVERSE EVENTS:
Arm/Group | DePuy Attune PS FB TKA
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes